CLINICAL TRIAL: NCT00246051
Title: Testing the Effectiveness of a Comprehensive Fatigue Management for the Police
Brief Title: Comprehensive Police Fatigue Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Charles Andrew Czeisler, MD, PhD, Charles A Czeisler, Ph.D., M.D.,, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: SL00067
Record Dates: First submitted 2005-09-13; First posted 2005-10-31 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Sleep Disorders; Sleep Apnea, Obstructive; Restless Legs Syndrome; Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders
Keywords: Police; Sleep; Fatigue; Work Hours; Sleep disorder; Performance
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea, Obstructive; Restless Legs Syndrome; Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Therapeutics

ARMS (3):
- Sleep Hygiene Education (Other)
  Interventions: Behavioral: Sleep Hygiene Education
- Expert-Led Sleep Disorders Screening and Treatment (Other)
  Interventions: Other: Expert-Led Sleep Disorders Screening and Treatment
- Online Sleep Disorders Screening (Other)
  Interventions: Other: Online Sleep Disorders Screening

INTERVENTIONS:
Behavioral: Sleep Hygiene Education — An education program, consisting of materials from experts in the field of fatigue management, will be provided to all police officers in the intervention group. Videotapes, slides, handouts and other educational material will be compiled to create a variety of information sources for police officers. Examples of materials to be incorporated into this training program would be the Operation Healthy Sleep Training Video, powerpoint created by the Harvard Work Hours, Health and Safety Group and pamphlets provided by the American Academy of Sleep Medicine.
  Arms: Sleep Hygiene Education
Other: Expert-Led Sleep Disorders Screening and Treatment — Expert-led sleep disorder screening and treatment will consist of visiting police stations and presenting an information session about Operation Healthy Sleep. The session will take place during work time. During the session, we will invite officers to take the Operation Healthy Sleep survey. All subjects that answer the survey indicating that they are at high risk on the Berlin Questionnaire will be contacted to arrange an initial appointment at our OSA research clinic. If they don't meet the criteria they will be disempanelled.
  1. Positive on the Berlin Questionnaire
  2. Clinic visit, exam with a physician, given a home diagnostic device (HDD)
  3. High risk on HDD, seen by physician, given a CPAP machine
  4. Follow up visit after 2-3 weeks, CPAP data downloaded and reviewed
  5. Contacted by a sleep health clinic at 3, 6, 12 months
  6. After 12 months subject will be referred to their primary care physician
  Arms: Expert-Led Sleep Disorders Screening and Treatment
Other: Online Sleep Disorders Screening — Online sleep disorder screening will be available to all police officers nation-wide through the Operation Healthy Sleep survey. All subjects that answer the survey questions indicating that they are at high risk of a sleep disorder will be notified either online following the completion of the survey or by email or a letter. Treatment and follow up will not be conducted for individuals who screen positive on the online version of the Operation Healthy Sleep survey.
  Arms: Online Sleep Disorders Screening

SUMMARY:
Police officers work some of the most demanding schedules known, which increases their risk of sleep deprivation and sleep disorders. The need to work frequent overnight shifts and long work weeks leads to acute and chronic partial sleep deprivation as well as misalignment of circadian phase. The public expects officers to perform flawlessly, but sleep deprivation and unrecognized sleep disorders significantly degrade cognition, alertness, reaction time and performance. In addition, both acute and chronic sleep deprivation adversely affect personal health, increasing the risk of gastrointestinal and heart disease, impairing glucose metabolism, and substantially increasing the risk of injury due to motor vehicle crashes.

We propose to conduct a randomized, prospective study of the effect on the safety, health, and performance of a police department of a Comprehensive Police Fatigue Management Program (CPFMP) consisting of the following interventions:

1. identification and treatment of police with sleep disorders;
2. caffeine re-education; and
3. initiation of a sleep, health and safety educational program.

These interventions were chosen because we believe them most likely to lead to measurable improvements on work hours, health, safety, and job performance, and because they are cost effective. The success of the CPFMP will be assessed through an experimental comparison with a standard treatment group that will receive sleep education in the absence of any accompanying interventions. The overall goal of our team will be sleep health detection and treatment program that can be disseminated to practitioners, policymakers and researchers nationwide to reduce police officer fatigue and stress; enhance the ability of officers to cope with shift schedules; improve the health, safety and performance of law enforcement officers; and thereby improve public safety.

ELIGIBILITY:
Inclusion Criteria:

* Active Sworn Police Officers

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2005-11; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Motor vehicle accidents as a function of miles traveled | 05/2005 - 07/2009
Number of on-the-job injuries | 05/2005 - 07/2009
Number of citations issued | 05/2005 - 07/2009
Number of arrests made | 05/2005 - 07/2009
Number of warnings issued | 05/2005 - 07/2009
Number of officer-initiated vehicle assists | 05/2005 - 07/2009
Number of sick leave days | 05/2005 - 07/2009
Sleep duration | 05/2005 - 07/2009
Sleep quality | 05/2005 - 07/2009
Alertness | 05/2005 - 07/2009
Performance | 05/2005 - 07/2009

SECONDARY OUTCOMES:
Job satisfaction | 05/2005 - 07/2009
Burnout | 05/2005 - 07/2009
Works hours | 05/2005 - 07/2009

CONTACTS AND LOCATIONS:
Overall Officials: Charles A. Czeisler, Ph.D., M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States